CLINICAL TRIAL: NCT05936411
Title: Study to Determine Interaction Patterns of Different Organs in Healthy Volunteers as a Basis for Better Patient Diagnostics Using PET/CT Imaging
Brief Title: Organ Interaction Patterns in Healthy Individuals for Improved PET/CT Diagnostics
Acronym: Healthy-PET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Univ.-Prof. Dr. Marcus Hacker, Head of the Division of Nuclear Medicine, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1707/2022
Record Dates: First submitted 2023-06-16; First posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-06

CONDITIONS: Healthy
Keywords: PET/CT; Total-Body PET/CT; Inter-Organ connection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Subjects (Other)
  Interventions: Device: Siemens Quadra PET/CT and [18F]FDG; Device: Apple i-Watch

INTERVENTIONS:
Device: Siemens Quadra PET/CT and [18F]FDG — The Siemens Quadra PET/CT, a clinically approved imaging device, is utilized in conjunction with the radiopharmaceutical tracer [18F]FDG in this study. The device allows for the acquisition of emission data across an extended axial field of view (axFOV) of 106 cm, covering an imaging range from the head to the thighs. The device's capabilities are leveraged to perform quantitative functional examinations of an extended axFOV. Subjects are scanned twice within a month for reproducibility standards. Each time, they are injected with 100MBq [18F]FDG and examined for 60 minutes in a dynamic scan. The tracer is used to build an atlas of normative glycolytic activities for most organs, excluding the brain. The glycolytic activities are measured as organ-based standardized uptake values. An ultra-low-dose CT scan is acquired to estimate mandatory attenuation correction factors.
Device: Apple i-Watch — The Apple i-Watch, a wearable smart device, is used to continuously monitor physiological signals from the subjects. These signals include heart rate, steps and distance, calories burned, sleep tracking, blood oxygen saturation (SpO2), electrocardiogram (ECG), and workout tracking. Subjects are required to wear the Apple i-Watch for three months prior to the first PET scan and up to three months after the second PET scan. The data collected from the Apple i-Watch is paired with the FDG-PET image readouts to identify relationships between lifestyle and glucose uptakes during the scan.

SUMMARY:
The study titled "Study to determine interaction patterns of different organs in healthy volunteers as a basis for better patient diagnostics using PET/CT imaging" is designed to investigate the interaction patterns of different organs in healthy volunteers. The information gathered is intended to be leveraged to enhance patient diagnostics using PET/CT imaging techniques.

DETAILED DESCRIPTION:
In the study titled "Study to determine interaction patterns of different organs in healthy volunteers as a basis for better patient diagnostics using PET/CT imaging," the investigators will utilize the Biograph Quadra from Siemens Healthineers. This clinically approved PET-based imaging platform enables the acquisition of emission data across an extended axial field of view (axFOV) of 106 cm.

The objective is to leverage the Quadra PET/CT's capabilities, which can perform quantitative functional examinations of an extended axFOV, large enough to cover an imaging range from the head to the thighs. This range is typically scanned in standard oncology re/staging scenarios using multiple, overlapping bed positions.

The aim is to convert the Quadra PET's higher volume sensitivity into a higher signal-to-noise ratio and image quality, and significantly reduce the injected radioactivity while maintaining the diagnostic quality of the PET images. Notably, all organs within the extended axFOV are covered synchronously by the PET measurement, allowing the examination of inter-organ signalling, a key factor in disease onset and progression.

It is understood that diseases like cancer cause deviations from normal inter-organ communication (homeostasis). To depict such deviations in the future, the aim is to establish a reference standard. This involves building a voxel-wise normative database of glycolytic activity across organs covered in the axFOV imaging range, which requires the acquisition of dynamic FDG-PET data of normal, disease-free individuals.

Additionally, the investigators seek to pair the FDG-PET image readouts with continuous physiological signals from an Apple i-watch wearable for identifying relationships between lifestyle and glucose uptakes during the scan. The objective is to build a normative database of voxel- and organ-based glycolytic uptake in 50 healthy volunteers. Subjects will be scanned twice for reproducibility standards and will wear a smartwatch for 3 months prior to the first PET scan and up to 3 months after the 2nd PET scan.

The hypothesis is that an atlas of normative glycolytic activities can be built with a test-retest variability of <15% (measured as organ-based standardized uptake value). The methodology involves using the Siemens Quadra PET/CT. Subjects come for test-retest within a month. Each time they will be injected 100MBq [18F]FDG and examined for 60 min (dynamic scan). An ultra-low-dose CT scan will be acquired to estimate mandatory attenuation correction factors.

No risks or adverse device effects are expected as the Quadra PET/CT is approved for clinical use.

ELIGIBILITY:
Inclusion Criteria:

- Adult subjects

Exclusion Criteria:

* Age < 18, common exclusion criteria for PET/CT scans
* known presence of cancer
* pregnancy or breastfeeding
* On-site blood glucose level > 150mg/dL
* Not able to lie still for 65 min

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Standardized Uptake Value (SUV) in gm/ml in Healthy Volunteers | 6 Months
  The primary outcome measure is the Standardized Uptake Value (SUV) in gm/ml, which is a measure of the image-derived radioactivity concentration and the whole body concentration of the injected radioactivity. The SUV will be reported as Mean and Standard Deviation. This measure will provide preliminary data about total body FDG perfusion and early biodistribution in a cohort of healthy volunteers. The SUV is calculated from the PET/CT scans using the Siemens Quadra PET/CT and [18F]FDG as the tracer.
Physiological Measurements from Apple i-Watch Wearable | 6 Months
  The secondary outcome measure is the physiological measurements collected from the Apple i-Watch wearable worn by the participants. These measurements include heart rate, steps and distance, calories burned, sleep tracking, blood oxygen saturation (SpO2),

IPD SHARING:
Plan to Share IPD: No